CLINICAL TRIAL: NCT03895385
Title: An Open-Label, Randomized, Parallel-Group, Single-Dose Study to Evaluate the Antibody Response of Influenza Vaccination Following Concomitant Exposure to Bimekizumab in Healthy Subjects
Brief Title: A Study to Evaluate the Antibody Response of Influenza Vaccination Following Concomitant Exposure to Bimekizumab in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Biopharma S.P.R.L. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UP0034
Record Dates: First submitted 2019-03-28; First posted 2019-03-29 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Healthy Volunteers
Keywords: BKZ; UCB4940; Healthy Subjects
MeSH Terms: interventions — bimekizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bimekizumab (Experimental): Subjects randomized to this arm will receive a single dose bimekizumab followed by inactivated influenza vaccine administered with a prefilled syringe at a predefined time point during the Treatment Period.
  Interventions: Drug: Bimekizumab
- No Treatment (No Intervention): Subjects randomized to this arm will receive the influenza vaccine administered with a prefilled syringe at a predefined time point during the Treatment Period.

INTERVENTIONS:
Drug: Bimekizumab — Subjects will receive a single dose bimekizumab at a predefined time point during the Treatment Period.
  Other Names: BKZ; UCB4940
  Arms: Bimekizumab

SUMMARY:
The purpose of the study is to evaluate whether administration of bimekizumab has an effect on the expected production of antibody titers to the influenza vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female aged ≥18 years and ≤55 years at the Screening Visit
* Subject must have a blood test with at least two influenza antibody titers ≤1/10 at the Screening Visit and have not developed any flu-like illness 2 weeks before the start of the study
* Female subjects of childbearing potential must not be lactating and have a negative serum pregnancy test at the Screening Visit, which is confirmed to be negative by urine testing prior to administration of bimekizumab. Female subjects of childbearing potential must agree to use a highly effective method of birth control during the study and for a period of 20 weeks after their last dose of the investigational medicinal product (IMP)
* Subject has a body weight of ≥45 kg and body mass index (BMI) between 18 and 32 kg/m2 (inclusive), at the Screening Visit

Exclusion Criteria:

* Subject has a known hypersensitivity to any excipients of bimekizumab
* Subject has a history of hypersensitivity to the influenza vaccine
* Subject is legally institutionalized or has a mental health condition or related care provision (eg, guardianship) that would impede the subject from providing voluntary informed consent to participate in the study
* Female subject who is pregnant, or plans to become pregnant during the study, or lactating, or sexually active with childbearing potential who is not using a medically accepted birth control method
* Male subjects who are planning a partner pregnancy during the study
* Subjects receiving vaccination of any kind within the 52 weeks prior to the Screening Visit or the influenza vaccination within 2 years prior to the Screening Visit. Live vaccines are not allowed during the study or for 20 weeks after the last dose of investigational medicinal product (IMP)
* Subject has a current or past history of gastrointestinal ulceration or other gastrointestinal disease, such as inflammatory bowel disease
* Subject has an active infection
* Subject has concurrent acute or chronic viral hepatitis B or C or human immunodeficiency virus (HIV) infection or human T-cell lymphotropic virus type-1 (HTLV-1)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2019-10-04 (Actual); Study Completion 2019-10-04 (Actual)

PRIMARY OUTCOMES:
Seroconversion response | From Baseline (Day 1 pre-dose) to 4 weeks post-vaccination (Day 43)
  A subject is considered as a seroconversion responder if the following is true: subject has either a pre-vaccination HI titer ≤1/10 and a 4-week post-vaccination HI titer ≥1/40 or a pre-vaccination HI titer >1/10 and a ≥4fold increase in HI titer 4 weeks after vaccination in at least 2 out of 4 serotypes.
Plasma concentration of bimekizumab (BKZ) | From Baseline (Day 1 pre-dose) at predefined time points (up to Day 140)
  Bimekizumab plasma concentrations by scheduled sampling time.
Incidence of Adverse Events (AE) from Baseline to Safety Follow Up | From Baseline to Safety Follow Up (up to Day 140)
  An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.

SECONDARY OUTCOMES:
Influenza antibody geometric mean titers (GMT) | From Baseline (Day 1 pre-dose) at predefined time points (up to Day 140)
  Post-vaccination influenza antibody geometric mean titers.
Area under the BKZ plasma concentration-time curve over the first 14 days AUC(0-14) | From Baseline (Day 1 pre-dose) at predefined time points (up to Day 14)
  The AUC(0-14) is the area under the plasma concentration-time curve from time zero to day 14.
Area under the BKZ plasma concentration-time curve over the first 28 days AUC(0-28) | From Baseline (Day 1 pre-dose) at predefined time points (up to Day 28)
  The AUC(0-28) is the area under the plasma concentration-time curve from time zero to day 28.
Area under the BKZ plasma concentration-time curve from time zero to last quantifiable concentration (AUCt) | From Baseline (Day 1 pre-dose) at predefined time points (up to Day 140)
  The AUCt is the area under the plasma concentration-time curve from time zero to last quantifiable concentration (AUCt) of BKZ as determined using the linear trapezoidal rule.
Area under the BKZ plasma concentration-time curve from time zero to infinity (AUC) | From Baseline (Day 1 pre-dose) at predefined time points (up to Day 140)
  The area under the plasma concentration-time curve from time zero to infinity (AUC) of BKZ is calculated as AUC=AUCt+Clast/λz, where Clast is the last quantifiable plasma concentration and λz is the apparent terminal elimination rate constant.
Maximum observed BKZ plasma drug concentration (Cmax) | From Baseline (Day 1 pre-dose) at predefined time points (up to Day 140)
  Cmax is the maximum plasma drug concentration of BKZ observed from pharmacokinetic samples taken at predefined time points.
Time of occurrence of the maximum observed BKZ plasma drug concentration (tmax) | From Baseline (Day 1 pre-dose) at predefined time points (up to Day 140)
  Tmax is the time to reach maximum plasma concentration.
Apparent terminal half-life (t1/2) | From Baseline (Day 1 pre-dose) at predefined time points (up to Day 140)
  Apparent terminal half-life, reported in units of days, as determined via simple linear regression (slope=-λz) of natural log (ln) concentration versus time for data points in the terminal phase of the concentration-time curve. t1/2 is calculated as ln2/λz.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (1):
- Up0034 001, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Due to the small sample size in this trial, IPD cannot be adequately anonymized i.e., there is a reasonable likelihood that individual participants could be re-identified. For this reason, data from this trial cannot be shared.